CLINICAL TRIAL: NCT00513110
Title: A Possible Therapeutic Role for Adenosine During Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: P.Pickkers MD PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007/099; CMO 2007/099
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2007-08

CONDITIONS: Endotoxemia
Keywords: Endotoxin; Adenosine; Caffeine; AMPD1 polymorphism
MeSH Terms: conditions — Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Endotoxin and AMPD1 polymorphism
  Interventions: Genetic: AMPD1 polymorphism
- 2 (Experimental): Endotoxin and intervention with caffeine
  Interventions: Drug: Caffeine infusion
- 3 (Placebo Comparator): Endotoxin combined with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Genetic: AMPD1 polymorphism — Endotoxin 2ng/kg to subjects with a AMPD1 polymorphism
  Arms: 1
Drug: Caffeine infusion — Endotoxin 2ng/kg combined with caffeine. Caffeine (4mg/kg) is used as an adenosine receptor antagonist.
  Arms: 2
Drug: placebo — Endotoxin 2ng/kg combined with saline infusion (0.9%)
  Arms: 3

SUMMARY:
The adenosine receptor is known for its anti-inflammatory actions and could therefore be a potential target in the treatment of sepsis and septic shock. Stimulation of the adenosine receptor could potentially lead to a decrease in inflammation and tissue damage.

Under normal conditions adenosine is formed either by an intracellular 5'nucleotidase, which dephosphorylates AMP, or by the hydrolysis of S-adenosylhomcysteine by hydrolase. An alternative pathway of AMP degradations is provided by the cytosolic enzyme AMP deaminase (AMPD), which catalyses the irreversible deamination of AMP to inosine monophosphate and ammonia.

In humans four AMPD isoforms have been described, named after the source from which they were initially purified; M (muscle), L (liver), E1 and E2 (erythrocyte), encoded by AMPD1, AMPD2 and AMPD3. Approximately 15-20% of Caucasian and African American individuals are heterozygous or homozygous for the 34C>T variant of AMPD1.

We hypothesize that healthy volunteers who have the polymorphism for AMPD1 have a less severe inflammatory response to LPS and show less (severe) organ failure. This hypothesis is based on the expected higher levels of adenosine in patients with the AMPD1 polymorphism. This hypothesis is strengthened by the fact that patients with coronary artery disease and the AMPD1 polymorphism show improved cardiovascular survival (Anderson JL et al. J Am Coll Cardiol 2000; 36: 1248-52) possibly based on higher adenosine levels by reduced AMPD activity. Furthermore the polymorphism predicts improved clinical outcome in patients with heart failure (Loh E et al. Circulation 1999) also based on a hypothetical elevation of adenosine.

We hypothesize that:

The C34T-polymorphism of the enzyme AMP-deaminase leads to a decreased inflammatory respons and thereby a decrease of LPS-induced tissue damage.

A second hypothesis is based on the antagonism of the adenosine receptor, by caffeine;

Antagonism of the adenosine receptor by caffeine leads to an increased LPS-induced inflammatory reaction and an increase in (subclinical) tissue damage?

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Drug-, nicotine-, alcohol abuses
* Tendency towards fainting
* Relevant medical history

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamics; heart rate variability | 24 hrs after LPS administration
Markers of Inflammation | 24 hrs after LPS administration
Cytokines | 24 hrs after LPS administration
Sensitivity to norepinephrine | 24 hrs after LPS administration
Endothelial-dependent and independent vasorelaxation | 24 hrs after LPS administration
Mediators of Vascular reactivity | 24 hrs after LPS administration
Markers of endothelial damage and circulating endothelial cells | 24 hrs after LPS administration
Urinary excretion of markers of renal injury | 24 hrs after LPS administration
Neurologic testing | 24 hrs after LPS administration
Adenosine and related nucleotide concentrations. | 24 hrs after LPS administration
Additional blood samples will be drawn for measurement of: TLR-expression, Genetics; micro array analyses and determination of intercellular signalling pathways. | 24 hrs after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD,PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Ramakers BP, Riksen NP, van den Broek P, Franke B, Peters WH, van der Hoeven JG, Smits P, Pickkers P. Circulating adenosine increases during human experimental endotoxemia but blockade of its receptor does not influence the immune response and subsequent organ injury. Crit Care. 2011;15(1):R3. doi: 10.1186/cc9400. Epub 2011 Jan 6. PMID 21211004
- [Derived] van den Boogaard M, Ramakers BP, van Alfen N, van der Werf SP, Fick WF, Hoedemaekers CW, Verbeek MM, Schoonhoven L, van der Hoeven JG, Pickkers P. Endotoxemia-induced inflammation and the effect on the human brain. Crit Care. 2010;14(3):R81. doi: 10.1186/cc9001. Epub 2010 May 5. PMID 20444270